CLINICAL TRIAL: NCT00510718
Title: A PHASE 1, OPEN-LABEL, DOSE-ESCALATION SAFETY AND PHARMACOKINETIC STUDY OF MDV3100 IN PATIENTS WITH CASTRATION-RESISTANT PROSTATE CANCER
Brief Title: A Phase 1 Study of MDV3100 in Patients With Castration-Resistant (Hormone-Refractory) Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: S-3100-1-01; C3431009 (Other: Alias Study Number); NCT00513812 (obsolete NCT alias)
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer; Hormone Refractory Prostate Cancer
Keywords: Prostate; Cancer; Hormone; Refractory; Castration
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MDV3100
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — MDV3100 daily until progression or dose-limiting toxicity
  Other Names: enzalutamide; Xtandi

SUMMARY:
This is a multi-center open-label dose-escalation study of a novel compound (MDV3100) to treat patients with castration-resistant (hormone-refractory) prostate cancer. Additional patients will be enrolled in expanded cohorts at doses determined to be tolerable. Patients who tolerate the drug and do not progress will be allowed to continue to look for PSA response.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, uncontrolled, dose-escalation study with dose-expansion at doses determined to be tolerated. Patients who tolerate the drug and do not progress will be allowed to continue treatment. The study endpoints are safety and tolerability and pharmacokinetics. PSA values will also be collected to look for PSA response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate;
2. Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration);
3. Progressive disease after medical or surgical castration,

Exclusion Criteria:

1. Metastases in the brain or active epidural disease. (Note: patients with treated epidural disease are allowed);

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2008-12-08 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MSKCC- Sidney Kimmel Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Investigational Pharmacy Services, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Gibbons JA, Ouatas T, Krauwinkel W, Ohtsu Y, van der Walt JS, Beddo V, de Vries M, Mordenti J. Clinical Pharmacokinetic Studies of Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1043-55. doi: 10.1007/s40262-015-0271-5. PMID 25917876
- [Derived] Scher HI, Beer TM, Higano CS, Anand A, Taplin ME, Efstathiou E, Rathkopf D, Shelkey J, Yu EY, Alumkal J, Hung D, Hirmand M, Seely L, Morris MJ, Danila DC, Humm J, Larson S, Fleisher M, Sawyers CL; Prostate Cancer Foundation/Department of Defense Prostate Cancer Clinical Trials Consortium. Antitumour activity of MDV3100 in castration-resistant prostate cancer: a phase 1-2 study. Lancet. 2010 Apr 24;375(9724):1437-46. doi: 10.1016/S0140-6736(10)60172-9. Epub 2010 Apr 14. PMID 20398925

RESULTS

PARTICIPANT FLOW:
Groups:
- MDV3100 (Enzalutamide): No Previous Chemotherapy: Participants with no prior exposure to chemotherapy received single oral dose of MDV3100 in 1 out of the 7 cohorts of 30, 60, 150, 240, 360, 480 or 600 milligram per day (mg/day) dose on Day 1 and were followed up for 6 days in single dose (dose escalation) period. Dose escalation from 30 to 600 mg/day continued until the maximum tolerated dose (MTD) was determined or until a dose of 600 mg/day was evaluated. After dose-escalation, the cohorts receiving 60-600 mg/day dose were expanded in multiple dose (dose expansion) period, where participants received MDV3100 according to their dose in single dose period for 84 days. This was followed by long-term dosing period in which participants continued to receive 160 mg/day dose of MDV3100 until withdrew of consent, dose limiting toxicity (DLT) or disease progression occurred. Participants were followed up for 30 days after last dose of study drug for safety follow up.
- MDV3100 (Enzalutamide): Post Chemotherapy: Participants with prior exposure to chemotherapy single oral dose of MDV3100 in 1 out of the 7 cohorts of 30, 60, 150, 240, 360, 480 or 600 mg/day dose on Day 1 and were followed up for 6 days in single dose (dose escalation) period. Dose escalation from 30 to 600 mg/day continued until the MTD was determined or until a dose of 600 mg/day was evaluated. After dose-escalation, the cohorts receiving 60-600 mg/day dose were expanded in multiple dose (dose expansion) period, where participants received MDV3100 according to their dose in single dose period, for 84 days. This was followed by long-term dosing period in which participants continued to receive 160 mg/day dose of MDV3100 until withdrew of consent, DLT or disease progression occurred. Participants were followed up for 30 days after last dose.
Period: Single Dose Period: 1 Week
Arm/Group | MDV3100 (Enzalutamide): No Previous Chemotherapy | MDV3100 (Enzalutamide): Post Chemotherapy
Started | 15 | 12
30 mg/Day | 3 | 0
60 mg/Day | 3 | 0
150/160 mg/Day | 2 | 1
240 mg/Day | 3 | 0
360 mg/Day | 4 | 2
480 mg/Day | 0 | 6
600 mg/Day | 0 | 3
Completed | 15 | 12
Not Completed | 0 | 0
Period: Multiple Dose Period: 12 Weeks
Arm/Group | MDV3100 (Enzalutamide): No Previous Chemotherapy | MDV3100 (Enzalutamide): Post Chemotherapy
Started | 65 (Participants who completed single dose period + new participants enrolled in multiple dose period.) | 75 (Participants who completed single dose period + new participants enrolled in multiple dose period.)
30 mg/Day | 3 | 0
60 mg/Day | 15 | 12
150/160 mg/Day | 15 | 13
240 mg/Day | 17 | 12
360 mg/Day | 15 | 13
480 mg/Day | 0 | 22
600 mg/Day | 0 | 3
Completed | 50 | 43
Not Completed | 15 | 32
Not completed — Adverse Event | 1 | 8
Not completed — PSA Disease Progression | 3 | 6
Not completed — Radiologic Disease Progression | 8 | 11
Not completed — Clinical Disease Progression | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- MDV3100 (Enzalutamide) 30 mg/Day: Participants received 30 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 60 mg /Day: Participants received 60 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 150/160 mg/Day: Participants who received 150 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period. This dose was then changed subsequently to 160 mg/day according to Protocol amendment. Participants continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 240 mg /Day: Participants received 240 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 360 mg /Day: Participants received 360 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 480 mg /Day: Participants received 480 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- MDV3100 (Enzalutamide) 600 mg /Day: Participants received 600 mg of Enzalutamide on Day 1 and were followed for 6 days in single dose period and continued to receive the same dose in multiple dose period for 84 days.
- Total: Total of all reporting groups
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day | Total
Number analyzed (Participants) | 3 | 27 | 28 | 29 | 28 | 22 | 3 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 15 | 10 | 8 | 10 | 7 | 3 | 54
  >=65 years | 2 | 12 | 18 | 21 | 18 | 15 | 0 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 27 | 28 | 29 | 28 | 22 | 3 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 3 | 24 | 28 | 27 | 27 | 22 | 3 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 4
  White | 3 | 26 | 28 | 28 | 25 | 22 | 3 | 135
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An adverse events (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 30 days after last dose of study treatment (approximately maximum of 129 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- MDV3100 (Enzalutamide) 160 mg /Day: Long Term Dosing Period: All participants after multiple dose period, continued to receive 160 mg/day oral dose of Enzalutamide in long term dosing period until they voluntarily withdrew, experienced a DLT or were diagnosed with disease progression.
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day | MDV3100 (Enzalutamide) 160 mg /Day: Long Term Dosing Period
Number analyzed (Participants) | 3 | 27 | 28 | 29 | 28 | 22 | 3 | 18
Participants | 0 | 6 | 14 | 8 | 6 | 1 | 1 | 10

2. Primary Outcome: Percentage of Participants With at Least 1 Dose-limiting Toxicity (DLT): Multiple Dose Period
Description: DLT was defined as a national cancer institute's common toxicity criteria for adverse events (NCI-CTCAE) version 3.0 grade 3 or greater toxicity regardless of perceived causality that is not improved by the use of adequate/maximal medical intervention. Grade 3 alopecia, fever without neutropenia, nausea, vomiting, fatigue, and self-limited or medically controllable adverse events were not considered as DLTs.
Time Frame: Baseline up to first 35 days of the study treatment in multiple dose period
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 27 | 28 | 29 | 28 | 22 | 3
percentage of participants | 0 | 0 | 0 | 0 | 1 | 1 | 2

3. Primary Outcome: Maximum Tolerated Dose (MTD) of MDV3100: Multiple Dose Period
Description: Tolerability was defined as if less than (<) 4/12 in participants with no prior exposure to MDV3100 (chemo-naive) and < 4/12 prior chemotherapy participants experienced a DLT within the first 35 days of the multiple dose period. For doses higher than 360 mg/day, tolerability was defined if <8/24 participants previously treated with chemotherapy experience a DLT within the first 35 days of the multiple dose period. MTD was defined as a dose below the intolerable dose.
Time Frame: Baseline up to first 35 days of the study treatment in multiple dose period
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: milligrams per day
Groups:
- MDV3100 (Enzalutamide) : All Participants: Participants received single oral dose of MDV3100 in 1 out of the 7 cohorts of 30, 60, 150, 240, 360, 480 or 600 mg/day dose on Day 1 and were followed up for 6 days in single dose (dose escalation) period. Dose escalation from 30 to 600 mg/day continued until the MTD was determined or until a dose of 600 mg/day was evaluated. After dose-escalation, the cohorts receiving 60-600 mg/day dose were expanded in multiple dose (dose expansion) period, where participants received MDV3100 according to their dose in single dose period for 84 days.
Arm/Group | MDV3100 (Enzalutamide) : All Participants
Number analyzed (Participants) | 140
milligrams per day | 240

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours Post Dose (AUC[0-24]) of MDV3100: Single Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24 hours post dose on Day 1 of Single Dose Period
Population: Pharmacokinetic (PK) evaluable population: all participants who received study drug and had sufficient PK samples for calculation of at least 1 MDV3100 PK parameter. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 0 | 0
microgram*hour per milliliter | 5.43 (11.80) | 15.64 (3.50) | 38.21 (23.64) | 58.39 (47.64) | 79.26 (19.29) |  |

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC[0-t]) of MDV3100: Single Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours postdose on Day 1 of Single Dose Period
Population: PK evaluable population: all participants who received study drug and had sufficient PK samples for calculation of at least 1 MDV3100 PK parameter. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 4 | 3
microgram*hour per milliliter | 21.2 (14.2) | 53.1 (4.1) | 145.3 (10.0) | 208.5 (44.0) | 320.2 (12.9) | 363.4 (38.7) | 391.9 (14.0)

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of MDV3100: Single Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3
microgram*hour per milliliter | 51.3 (39.8) | 92.7 (19.0) | 331.5 (14.6) | 459.2 (32.7) | 706.7 (17.7) | 952.7 (42.4) | 865.0 (34.6)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MDV3100: Single Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: PK evaluable population: all participants who received study drug and had sufficient PK samples for calculation of at least 1 MDV3100 PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3
hours | 1.98 [0.42 to 4.00] | 0.50 [0.48 to 1.00] | 0.53 [0.50 to 1.98] | 1.00 [0.57 to 1.00] | 1.03 [0.53 to 2.20] | 1.54 [0.53 to 2.08] | 1.03 [1.03 to 2.00]

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MDV3100: Single Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3
microgram per milliliter | 0.43 (15.97) | 1.65 (28.77) | 3.30 (22.85) | 5.19 (18.64) | 6.68 (39.61) | 5.93 (66.03) | 5.17 (19.51)

9. Secondary Outcome: Apparent Terminal Elimination Half-Life (T1/2) of MDV3100: Single Dose Period
Description: T 1/2 is the time measured for the plasma concentration of MDV3100 to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3
hours | 164.9 (69.8) | 100.5 (30.9) | 143.7 (34.8) | 138.9 (22.6) | 149.1 (26.1) | 144.0 (68.4) | 130.4 (37.7)

10. Secondary Outcome: Apparent Volume of Distribution (V/F) of MDV3100: Single Dose Period
Description: Volume of distribution is defined as the theoretical volume in which the total amount of MDV3100 would need to be uniformly distributed to produce the desired plasma concentration of MDV3100. Apparent volume of distribution after oral dose (V/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3
liters | 131.7 (15.6) | 90.5 (16.0) | 91.89 (13.31) | 103.8 (48.5) | 108.2 (15.8) | 97.4 (30.7) | 126.4 (8.8)

11. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of MDV3100: Single Dose Period
Description: Clearance of a MDV3100 is a measure of the rate at which a MDV3100 is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 120 hours post dose on Day 1 of Single Dose Period
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3
liters per hour | 0.585 (39.810) | 0.647 (18.988) | 0.453 (14.583) | 0.523 (32.679) | 0.509 (17.711) | 0.504 (42.437) | 0.694 (34.625)

12. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours Post Dose (AUC[0-24]) of MDV3100: Multiple Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 24 hours post dose on Day 84 of Multiple Dose Period
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 20 | 22 | 29 | 14 | 1 | 0
microgram*hour per milliliter | 60.0 (21.0) | 109.8 (34.4) | 291.7 (24.9) | 395.7 (27.4) | 488.9 (23.9) | 463.1 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. |

13. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MDV3100: Multiple Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 24 hours post dose on Day 84 of Multiple Dose Period
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 21 | 23 | 29 | 16 | 1 | 0
hours | 2.07 [1.00 to 3.92] | 1.07 [0.50 to 23.67] | 1.00 [0.00 to 25.80] | 1.08 [0.00 to 26.17] | 1.57 [0.48 to 24.08] | 0.00 [0.00 to 0.00] |

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MDV3100: Multiple Dose Period
Time Frame: Pre-dose, 0.5, 1, 2, 24 hours post dose on Day 84 of Multiple Dose Period
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 21 | 23 | 29 | 16 | 1 | 0
microgram per milliliter | 2.76 (21.10) | 5.49 (28.88) | 14.07 (25.36) | 18.91 (26.57) | 24.57 (21.00) | 27.90 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. |

15. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of MDV3100: Multiple Dose Period
Time Frame: Pre-dose on Day 1 of Multiple Dose Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 22 | 24 | 25 | 21 | 16 | 3
microgram per milliliter | 0.10 (0.03) | 0.00 (0.00) | 0.04 (0.19) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 1.89 (0.55)

16. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of MDV3100: Multiple Dose Period
Description: as for outcome 11
Time Frame: Pre-dose, 0.5, 1, 2, 24 hours post dose on Day 84 of Multiple Dose Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 20 | 22 | 29 | 14 | 1 | 0
liters per hour | 0.507 (0.111) | 0.580 (0.245) | 0.530 (0.149) | 0.628 (0.179) | 0.755 (0.176) | 1.037 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. |

17. Other Pre Specified Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response at Day 84: Multiple Dose Period
Description: Prostate-specific antigen is a glycoprotein considered as a biomarker for the response to therapy in men with prostate cancer. A 50 percent (%) decline in PSA from baseline to the PSA level at Day 84 was considered as a PSA response.
Time Frame: Baseline, Day 84
Population: Analysis population included all enrolled participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day
Number analyzed (Participants) | 3 | 24 | 24 | 20 | 21 | 11 | 0
percentage of participants | 33.3 [0.8 to 90.6] | 50.0 [29.1 to 70.9] | 66.7 [44.7 to 84.4] | 75.0 [50.9 to 91.3] | 71.4 [47.8 to 88.7] | 45.5 [16.7 to 76.6] |

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study treatment (approximately maximum of 129 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or participant may have experienced both SAE and NSAE. Analysis population included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | MDV3100 (Enzalutamide) 30 mg/Day | MDV3100 (Enzalutamide) 60 mg /Day | MDV3100 (Enzalutamide) 150/160 mg/Day | MDV3100 (Enzalutamide) 240 mg /Day | MDV3100 (Enzalutamide) 360 mg /Day | MDV3100 (Enzalutamide) 480 mg /Day | MDV3100 (Enzalutamide) 600 mg /Day | MDV3100 (Enzalutamide) 160 mg /Day: Long Term Dosing Period
Serious Adverse Events (participants affected / at risk) | 0/3 | 6/27 | 14/28 | 8/29 | 6/28 | 1/22 | 1/3 | 10/18
Other Adverse Events (participants affected / at risk) | 3/3 | 27/27 | 27/28 | 29/29 | 28/28 | 21/22 | 3/3 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDV3100 (Enzalutamide) 30 mg/Day (N=3) | MDV3100 (Enzalutamide) 60 mg /Day (N=27) | MDV3100 (Enzalutamide) 150/160 mg/Day (N=28) | MDV3100 (Enzalutamide) 240 mg /Day (N=29) | MDV3100 (Enzalutamide) 360 mg /Day (N=28) | MDV3100 (Enzalutamide) 480 mg /Day (N=22) | MDV3100 (Enzalutamide) 600 mg /Day (N=3) | MDV3100 (Enzalutamide) 160 mg /Day: Long Term Dosing Period (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDV3100 (Enzalutamide) 30 mg/Day (N=3) | MDV3100 (Enzalutamide) 60 mg /Day (N=27) | MDV3100 (Enzalutamide) 150/160 mg/Day (N=28) | MDV3100 (Enzalutamide) 240 mg /Day (N=29) | MDV3100 (Enzalutamide) 360 mg /Day (N=28) | MDV3100 (Enzalutamide) 480 mg /Day (N=22) | MDV3100 (Enzalutamide) 600 mg /Day (N=3) | MDV3100 (Enzalutamide) 160 mg /Day: Long Term Dosing Period (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 3 | 4 | 3 | 2 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Vision blurred (Eye disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 4 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 10 | 8 | 7 | 11 | 6 | 1 | 6
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 8 | 3 | 4 | 9 | 1 | 8
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5 | 3 | 1 | 6 | 4 | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 3 | 4 | 5 | 3 | 4 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 3 | 3 | 2 | 3 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 17 | 19 | 20 | 23 | 16 | 1 | 13
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 3 | 3 | 3 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Oedema peripheral (General disorders) | 1 | 6 | 9 | 5 | 6 | 1 | 0 | 3
Pain (General disorders) | 0 | 4 | 2 | 3 | 3 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 4 | 4 | 2 | 1 | 2 | 1 | 1
Sluggishness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Axillary candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blastocystis infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 4 | 4 | 1 | 2 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 4 | 1 | 3 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunoglobulins increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Light chain analysis increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 6 | 1 | 2 | 1 | 3 | 0 | 1
Weight increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 6 | 8 | 4 | 9 | 4 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6 | 3 | 5 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 11 | 8 | 7 | 8 | 5 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 11 | 5 | 8 | 9 | 6 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 5 | 2 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 2 | 5 | 5 | 4 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 1 | 1 | 1 | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 9 | 6 | 9 | 6 | 3 | 0 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 3 | 1 | 1 | 4 | 4 | 1 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 7 | 5 | 7 | 4 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 5 | 3 | 8 | 3 | 0 | 1
Headache (Nervous system disorders) | 0 | 6 | 2 | 6 | 5 | 5 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 3 | 2 | 1 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Judgement impaired (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 3 | 1 | 1 | 3 | 0 | 2
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Mental retardation severity unspecified (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 3 | 1 | 3 | 0 | 2 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 5
Restless legs syndrome (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Vertigo positional (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 2 | 0 | 3 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1 | 4 | 0 | 0
Impatience (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 5 | 2 | 2 | 5 | 1 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phobia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 4 | 1 | 4 | 1 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 5 | 2 | 1 | 5 | 1 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 4 | 2 | 3 | 0 | 0 | 6
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 5 | 7 | 3 | 2 | 0 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 7 | 10 | 6 | 3 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 4 | 2 | 1 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 7 | 7 | 2 | 6 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2 | 2 | 3 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrophy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 2
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Schamberg's disease (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ectropion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Glare (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Refraction disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 5 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecal volume decreased (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip exfoliation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 11 | 6 | 19 | 11 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus ani (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.